CLINICAL TRIAL: NCT02969746
Title: Activates Charcoal for Patients Undergoing Invasive Procedure Delayed Due to Direct Oral Anticoagulants
Acronym: CACAOD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Feasibility issues, difficulties in the patient pathway, advances in knowledge
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACAOD
Record Dates: First submitted 2016-11-09; First posted 2016-11-21 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Anticoagulants; Circulating, Hemorrhagic Disorder
Keywords: activated charcoal, direct oral anticoagulant
MeSH Terms: conditions — Hemorrhagic Disorders; Anthrax | interventions — Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Charcoal (Experimental): Patients will receive a single dose (20 gram) of oral activated charcoal
  Interventions: Drug: Activated Charcoal
- control (No Intervention): Standard practice

INTERVENTIONS:
Drug: Activated Charcoal — Patients will take oral activated charcoal after randomization in the intervention arm.
  A blood sample(TO) will be collected after patient enrollment and before charcoal administration and 4 blood samples will be collected on a 8h length period (T1 to T4)
  Arms: Charcoal

SUMMARY:
This is a prospective, multicentric, randomized, open labeled superiority trial

This study aims to evaluate the efficacy of oral activated charcoal for improving elimination of direct oral anticoagulants ( Rivaroxaban, Apixaban) in case of an unscheduled invasive procedure delayed to this anticoagulant treatment.

The primary outcome is the anticoagulant's half life. Plasma concentration will be measured by liquid chromatography-mass spectrometry for the main analysis (pharmacokinetic).

A total of 140 patients will randomly be assigned to the charcoal or control group, stratified according to their anticoagulant drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients under direct oral anticoagulant treatment (Apixaban, Rivaroxaban or Dabigatran)
* Age ≥18 years;
* Clinical condition needing a surgery or invasive procedure ( lumbar puncture, biopsy...), needing anticoagulant treatment interruption and intervention to be postponed
* Signed informed consent

Exclusion Criteria:

* Urgent immediate surgery without any possibility to wait for 24 hours
* contraindication for receiving oral treatment
* Active uncontrolled bleeding or bleeding in critical organ
* Hemodynamic instability, shock
* Known anticoagulant concentration < 50ng/mL
* drug intoxication
* Fructose intolerance, glucose and galactose malabsorption syndrome, sucrase-isomaltase deficit
* Treated epileptic disease
* Pregnant or breast feeding
* Patient under guardianship
* No insurance cover
* Patient unable to give his consent
* Participation to another therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Direct Oral Anticoagulant half life | 0 to 8 hours

SECONDARY OUTCOMES:
Time to obtain a plasmatic concentration lower than 50ng/mL | 0 to 8 hours
Rate of bleeding and/or thromboembolic complications after activated charcoal administration or not. | until Day 7
Number of patients with adverse events. | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Moumneh, Dr, Principal Investigator — Sponsor GmbH
Locations (5):
- France (5):
  - Chu Angers, Angers
  - CHU Clermont-ferrand, Cléron
  - CH Le MANS, Le Mans
  - CHU de Poitiers, Poitiers
  - CHU de St Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No